CLINICAL TRIAL: NCT02656836
Title: Home Tonometry for Monitoring Glaucoma:a Pilot Study of the Icare Home Tonometer
Brief Title: Home Tonometry With the I-care Tonometer for Glaucoma
Status: Completed | Type: Observational
Sponsor: Queen's University, Belfast (Other)
Collaborators: Belfast Health and Social Care Trust (Other)
Responsible Party: Principal Investigator, Professor Augusto Azuara-Blanco, Professor, Queen's University, Belfast
Other Study IDs: REC 15/EM/0217
Record Dates: First submitted 2016-01-11; First posted 2016-01-15 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Home tonometry, diagnostic study — Evaluating intraocular pressure
  Other Names: I-care tonometer

SUMMARY:
The overall objective of the study is to scope the self-management for self-monitoring glaucoma using home tonometry.

DETAILED DESCRIPTION:
Monitoring of glaucoma requires frequent evaluation of IOP and disease severity, typically with visual field tests. When a patient is diagnosed with glaucoma an optimum level of IOP (or target IOP) is determined based on patient's characteristics, such as severity of disease and life expectancy. In current models of care patients have their IOP measured at the clinic at different intervals. If the IOP is noted to be high, or above the patient's target, additional treatment is recommended. Accurate and frequent IOP measurements at different points in time are thus imperative.

Tonometry is usually conducted by clinicians in an eye clinic. Some tonometers (e.g., Icare) have the potential to be used by the individual for home monitoring of IOP for patients with suspected glaucoma/glaucoma. Self-monitoring of IOP via home tonometry will allow patients to undergo IOP measurements at different points in time (e.g., early morning and night-time, and it can help determine diurnal changes and spikes).

The overall objective of the current study is to conduct a feasibility pilot study on the home tonometer (Icare), acquiring initial experience with the Icare tonometer. For this purpose investigators will train up to 20 individuals on how to use the device. Investigators will ask them to record in a diary their IOP twice a day for a period of 2 weeks. Investigators will then compare IOP outcomes with the measurement taken at the clinic. Patients and clinicians will be masked to the IOP data.

ELIGIBILITY:
Inclusion Criteria:

1. Attending the glaucoma clinic for monitoring (for glaucoma or ocular hypertension)
2. Aged 18 years or over
3. Patient deemed able to monitor their IOP at home (by themselves or a helper)

Exclusion Criteria:

1. Not receiving IOP monitoring (for glaucoma or ocular hypertension)
2. Aged <18 years
3. Patients deemed unable to monitor their IOP at home (and do not have someone who can help them) e.g., apparent physical or cognitive impairments that will not allow for the use of a home tonometer
4. Had surgery for their glaucoma (glaucoma surgery only; other surgeries included e.g., cataract surgery)
5. Patient has preexisting corneal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with glaucoma attending clinic
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Augusto Azuara-Blanco, Principal Investigator — Queen's University, Belfast
Locations (1):
- Centre for Experimental Medicine QUB, Belfast, Co.Antrim, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Could not recruit target number of participants within the time frame
Groups:
- Home Tonometry Group: No comparator
Period: Overall Study
Arm/Group | Home Tonometry Group
Started | 9
Completed | 6
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Home Tonometry Group
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure
Description: Intraocular pressure in mmHg units, obtained by tonometers. The investigators will determine agreement of intraocular pressure (IOP) measured using the home tonometer (patient) compared with IOP measured in the clinic.
Time Frame: Two weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Home Tonometry Group
Number analyzed (Participants) | 6
mmHg | -1.85 (3.95)

2. Secondary Outcome: Proportion of Patients Able and Willing to Use the Tonometer
Description: Proportion of patients willing to use the tonometer but are unable to. Patient feedback reported via questionnaire
Time Frame: Two weeks
Reporting Status: Not Posted

3. Secondary Outcome: Proportion of Patients With an Adverse Event
Description: Any adverse event or complication associated with the use of the device. Expected side effects will be corneal erosion, and ocular irritation.
Time Frame: One month
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Home Tonometry Group
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes